CLINICAL TRIAL: NCT06153589
Title: Effectiveness of Musicotherapy in Reducing Pain Induced by Leg Ulcer Care: a Randomized, Controlled, Open-label, Parallel-arm Study
Brief Title: Effectiveness of Musicotherapy in Reducing Pain Induced by Leg Ulcer Care
Acronym: MUS-ICAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Music Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23_RIPH2-10
Record Dates: First submitted 2023-11-13; First posted 2023-12-01 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Debridement Care; Leg Ulcer; Leg Ulcers Venous; Pain
Keywords: Debridement; Venous leg ulcer; Pain
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Musicotherapy + debridement and usual analgesic protocol (Experimental): Patients in the experimental arm will receive classic debridement care and usual use of analgesic treatment, accompanied by a musicotherapy session respecting the standardized method of the U-shaped sequence.
  Interventions: Other: Musicotherapy
- Debridement and usual analgesic protocol (No Intervention): Patients in the experimental arm will receive classic debridement care and usual use of analgesic treatment.

INTERVENTIONS:
Other: Musicotherapy — Musicotherapy will be offered to patients who meet the eligibility criteria, and have been randomized to the experimental arm.
  Patients will only be seen once during the study. Patients are placed in individual rooms. Hifi audio headphones (equipped with hygienic earcups) and a tablet equipped with the Music Care application will be offered to patients in the experimental group and the investigators will help them choose the style of music, which respects the U-shaped sequence.
  The Music Care application has proven that the use of headphones allows the patient to be isolated and therefore to obtain less parasitic care. He will be told at the start of the session that he can ask to interrupt it if he wishes to communicate with the team, particularly regarding possible pain.
  The musicotherapy session begins before the act of debridement (10 minutes before), lasts during the act (40 minutes maximum), and continues for 10 minutes after the end of the debridement.
  Arms: Musicotherapy + debridement and usual analgesic protocol

SUMMARY:
Venous leg ulcer is the final stage of chronic venous disease and only develops due to advanced chronic venous insufficiency. The problems caused by venous disease are initially minor and often neglected, but can impact the quality of life of patients.

The prevalence of leg ulcers is estimated at 1% of the general population and 3% to 5% of subjects over 65 years old. Its prevalence increases with age in both men and women.

Managing chronic ulcers requires a certain number of care procedures, including debridement.

The act of treatment by mechanical debridement is little relieved by the analgesics given beforehand, and can be painful, with risks of bleeding.

Musicotherapy, particularly the U-shaped method, has shown its effectiveness in the treatment of pain and anxiety in several areas (geriatrics, intensive care, rheumatology, oncology, etc.).

The standardized musicotherapy method of the U-shaped sequence was developed and initially evaluated by clinical studies coordinated by the INSERM unit U1061 (Pr. Jacques Touchon; Dr. Stéphane Guétin).

Following the publication of numerous controlled, randomized studies presenting results on the effectiveness in the treatment of pain and anxiety, a digital application was developed in order to standardize the method. The Music Care health application is now a Class 1 Medical Device, with CE marking obtained.

This "U-shaped sequence" is standardized and has been clinically validated, which makes Music Care a unique tool available for pain relief.

No studies have been found in the literature regarding the use of music therapy during debridement care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient,
* Patient followed at the M@diCICAT healing center requiring wound debridement :

  * For a venous or arterial ulcer or necrotizing angiodermatitis of the lower limbs,
  * Having the ability to verbalize about their pain (communicating),
  * With a planned debridement time of less than 40 minutes.
* Patient affiliated to or beneficiary of a social security scheme,
* Patient having given free, informed and express consent.

Exclusion Criteria:

* Patient with a diabetic foot (loss of sensitivity-neuropathy),
* Patient not requiring a debridement session,
* Patient with an infected ulcer (abscess, etc.),
* Patient with critical ischemia,
* Patient with hearing problems,
* Patient with cognitive disorders,
* Patient placed under legal protection, guardianship or curatorship,
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of "U" musicotherapy in the management of pain induced by debridement in patients with chronic wounds of the lower limb | 18 months
  Variation in physical pain assessed by VAS (Visual Analogue Scale from 0 to 10)

SECONDARY OUTCOMES:
To evaluate the effectiveness of "U" music therapy in reducing the consumption of analgesics during and after debridement treatment on a chronic wound of the lower limb. | 18 months
  Consumption of analgesics during and after debridement (Level 1-2 or 3, route, dosage, frequency).
To evaluate the effectiveness of "U" music therapy in the variation of anxiety induced by debridement in patients with chronic wounds of the lower limb. | 18 months
  Variation in anxiety according to the VAS anxiety scale, (VAS anxiety 10 min after debridement) - (VAS anxiety 10 min before debridement). The anxiety VAS will be collected at the two times according to the patient's assessment.
To evaluate the variation of blood pressure before and after debridement treatment on a chronic wound of the lower limb. | 18 months
  Blood pressure variation before and after debridement.
To evaluate the variation of heart rate before and after debridement treatment on a chronic wound of the lower limb. | 18 months
  Heart rate variation before and after debridement.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Guitteaud, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No